CLINICAL TRIAL: NCT04088682
Title: Clinical Performance and Quality Measures for Adults With Acute ST-Elevation Myocardial Infarction in China
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: NCCQI-CAD
Record Dates: First submitted 2019-09-09; First posted 2019-09-13 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: clinical performance; quality measures; ST-Elevation myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All hospitals: All hospitals will take the treatment quality improvement strategies and tools into implementation.
  Intervention: Behavioral: Quality improvement strategies and tools
  Interventions: Behavioral: Quality improvement strategies and tools

INTERVENTIONS:
Behavioral: Quality improvement strategies and tools — Quality improvement strategies and tools

SUMMARY:
This study aims to investigate and evaluate clinical performance and quality measures for adults with acute ST-elevation myocardial infarction (STEMI) in China. Further more, the investigates like to develop quality improvement strategies and relevant tools focusing on treatment and clinical outcome in patients with STEMI. This is a annually survey , through consecutively recruiting all eligible inpatients and collecting relevant medical information, the performance of all participating hospitals. Further, quality improvement strategies including summary of clinical performance and quality measures, clinical pathways and team building will be organized for the purpose of quality improvement. All hospitals will consecutively recruit qualified patients in the same method adopted in baseline period. Then the reperfusion rates and other performance measures will be compared annually.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a major concern in public health globally, as well as in China, and remarkable variations of resources available and health system performance have been noted. Acute myocardial infarction is one of the leading causes of mortality and morbidity, both in rural and urban area.

This study aims to investigate and evaluate clinical performance and quality measures for adults with acute ST-elevation myocardial infarction (STEMI) in China. Further more, the investigates like to develop quality improvement strategies and relevant tools focusing on treatment and clinical outcome in patients with STEMI.

This is a annually survey , through consecutively recruiting all eligible inpatients and collecting relevant medical information, the performance of all participating hospitals. Demographic characteristics, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be obtained and then, the treatment pattern and outcomes will be evaluated. Further, quality improvement strategies including summary of clinical performance and quality measures, clinical pathways and professional training will be organized for the purpose of quality improvement. All hospitals will consecutively recruit qualified patients in the same method adopted in baseline period. Then the reperfusion rates and other performance measures will be compared annually.

New knowledge will be generated about STEMI management in China, to improve STEMI patients prognosis in future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI who arrive at the hospital within 48 hours from the symptoms onset.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with STEMI who arrive at the hospital within 48 hours from the symptoms onset
Sampling Method: Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Aspirin at arrival | 24 hours after admission
  Proportion of aspirin use within 24 hours of admission among eligible patients
Clopidogrel (or ticagrelor) at arrival | 24 hours after admission
  Proportion of Clopidogrel (or ticagrelor) use within 24 hours of admission among eligible patients
β-blockers at arrival | 24 hours after admission
  Proportion of β-blockers use within 24 hours of admission among eligible patients
ECG at arrival | 24 hours after admission
  Proportion of ECG test within 10 minutes of admission among eligible patients
Reperfusion therapy rate | 24 hours after admission
  Reperfusion therapy rate is defined as utilization rate of thrombolytic therapy or primary PCI treatment among patients indicated with the reperfusion therapy.
Time delay from failure of fibrinolysis to angiography(The time from start of fibrinolysis to evaluation of its efficacy is 60-90min) | 10 days on average (during hospitalization)
  The proportion of failure of fibrinolysis to balloon within 90 minutes among all patients receiving PCI.
Time delay from start of fibrinolysis to angiography(if fibrinolysis is successful) | 10 days on average (during hospitalization)
  The proportion of from fibrinolysis to balloon (if fibrinolysis is successful) within 2-24hours among all patients receiving PCI.
Timeliness of thrombolytic therapy | 24 hours after admission
  The proportion of door to needle time (D2N) within 30 minutes among all patients receiving fibrinolytic therapy.
Timeliness of primary PCI | 24 hours after admission
  The proportion of door to balloon (D2B) within 90 minutes among all patients receiving primary PCI.
Door-in-Door-Out Time | 24 hours after admission
  Percentage of patients whose median time from the emergency department arrival at STEMI referral facility to emergency department discharge from STEMI referral facility is equal or less than 30 min. discharge from STEMI referral facility is 30 min.
Time to Primary PCI Among Transferred Patients | 24 hours after admission
  Percentage of patients whose median time from first medical contact (at or before emergency department arrival to the STEMI referral facility [e.g., non-PCI-capable facility]) to primary PCI at the STEMI receiving facility (PCI-capable facility) is equal or less than 120 min
Evaluation of LDL-C | 10 days on average (during hospitalization)
  Percentage of patients with documentation in the hospital record that LDL-C is evaluated during hospitalization
Evaluation of left ventricular ejection fraction | 10 days on average (during hospitalization)
  Percentage of patients with documentation in the hospital record that left ventricular ejection fraction is evaluated during hospitalization
Aspirin use during hospitalization | 10 days on average (during hospitalization)
  Proportion of Aspirin use during hospitalization among eligible patients.
Clopidogrel (or ticagrelor) use during hospitalization | 10 days on average (during hospitalization)
  Proportion of Clopidogrel (or ticagrelor) use during hospitalization among eligible patients.
β-blockers use during hospitalization | 10 days on average (during hospitalization)
  Proportion of β-blockers use during hospitalization among eligible patients.
Angiotensin-converting enzyme inhibitor /angiotensin II receptor blocker use during hospitalization | 10 days on average (during hospitalization)
  Proportion of Angiotensin-converting enzyme inhibitor /angiotensin II receptor blocker use during hospitalization among eligible patients.
Statins use during hospitalization | 10 days on average (during hospitalization)
  Proportion of statins use during hospitalization among eligible patients.
Aspirin use at discharge | 10 days on average (during hospitalization)
  Proportion of aspirin use at discharge among eligible patients.
Clopidogrel (or ticagrelor) use at discharge | 10 days on average (during hospitalization)
  Proportion of Clopidogrel (or ticagrelor) use at discharge among eligible patients.
β-blockers use at discharge | 10 days on average (during hospitalization)
  Proportion of β-blockers use at discharge among eligible patients.
angiotensin-converting enzyme inhibitor /angiotensin II receptor blocker use at discharge | 10 days on average (during hospitalization)
  Proportion of angiotensin-converting enzyme inhibitor /angiotensin II receptor blocker use at discharge among eligible patients.
Statins use at discharge | 10 days on average (during hospitalization)
  Proportion of statins use at discharge among eligible patients.
Aldosterone Antagonist at Discharge | 10 days on average (during hospitalization)
  Proportion of Aldosterone Antagonist use at discharge among eligible patients.
Smoking cessation advice/ counseling at Discharge | 10 days on average (during hospitalization)
  Proportion of patients received smoking cessation advice/ counseling
all-cause mortality during hospitalization | 10 days on average (during hospitalization)
  Proportion of patients who were all-cause death during hospitalization
Cardiac mortality during hospitalization | 10 days on average (during hospitalization)
  Proportion of patients who were cardiac death during hospitalization
30-day all-cause mortality | From admission to 30days
  Proportion of patients who were all-cause death from admission to 30days
30-day cardiac mortality | From admission to 30days
  Proportion of patients who were cardiac death from admission to 30days
30-day readmission rates | From hospital discharge to 30 days
  Proportion of patients readmission from hospital discharge to 30days
Cost during hospitalization | 10 days on average (during hospitalization)
  Cost during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Hongjian Wang, Beijing, Beijing Municipality, China